CLINICAL TRIAL: NCT05988996
Title: Peer Support for Black and Latino Families With an Infant in the NICU
Brief Title: Peer Support Groups for Families With an Infant in the NICU
Status: Enrolling by invitation | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Legacy Health System (Other); Providence Health & Services (Other)
Responsible Party: Principal Investigator, Sasha Ondusko, Principal Investigator, Oregon Health and Science University
Other Study IDs: STUDY00025682
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Stress
Keywords: Parental stress; Parental anxiety; NICU; Peer support
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- African American and Black: One cohort includes families that identify as Black, African American, or African attending the racially concordant peer group sessions.
  Interventions: Behavioral: Participant guided peer support gathering
- Latino English Preferred: One cohort includes families that identify as Latino, Hispanic, Chicano and language preference of English attending the ethnically concordant peer group sessions.
  Interventions: Behavioral: Participant guided peer support gathering
- Latino Spanish preferred: One cohort includes families that identify as Latino, Hispanic, Chicano and language preference of Spanish attending the ethnically and linguistically concordant peer group sessions.
  Interventions: Behavioral: Participant guided peer support gathering

INTERVENTIONS:
Behavioral: Participant guided peer support gathering — This prospective observational cohort study will be assessing parental stress, anxiety, and sense of belonging before and after participant attendance at the culturally concordant peer group session.

SUMMARY:
The goal of this observational study is to learn the impact of race, ethnicity, and language matched peer support groups on parental stress, anxiety, and sense of belonging for families who have or have had an infant hospitalized in the Neonatal Intensive Care Unit (NICU). The main questions aim to answer: Do race, ethnicity, and language matched peer support groups decrease parental stress and anxiety and improve sense of belonging of parents while their baby is hospitalized in the NICU? And, are there any changes that should be made to the format of the peer support group sessions?

Participants will be invited to attend a peer support group that is matched for race, ethnicity, and language. Participants will have the option of filling out a survey on stress, anxiety, and sense of belonging before and after the peer group session. Additionally, participants will have the option of filling out a satisfaction survey after the peer group session.

DETAILED DESCRIPTION:
The study will be observational research wherein participants who want to attend a peer support group, will have the option of filling out surveys before and after peer support group attendance. Surveys are voluntary and the only way of assessing the behavioral outcome (impact on parental stress, anxiety, and sense of belonging); families can attend the peer support groups even if the family member does not want to participate in the survey.

ELIGIBILITY:
Inclusion Criteria:

* Parental or guardian self-identified as Black, African American, African, Latino, Hispanic, Chicano
* Parent or guardian of infant that was or is admitted to Oregon Health & Science University, Randall Children's Hospital, or Providence Health NICU in Portland, OR

Exclusion Criteria:

* Parent or guardian age less than 18 years old
* Preferred language other than English or Spanish (including if preferred communication is sign language)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from the population of people who are attending the peer support group sessions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Parental stress | 1 week prior to 2 days after peer group session
  The degree of parental stress in the NICU will be assessed using the Parental Stressor Scale: Neonatal Intensive Care Unit validated tool. The minimum and maximum values are 26 and 130 respectively, with higher scores indicating higher parental stress.

SECONDARY OUTCOMES:
Parental sense of belonging | 2 days after peer group session
  Sense of belonging will be assessed with three non-validated questions about community and within NICU sense of belonging questions. The scoring system is a 5-point Likert scale with an option for "Not Applicable". The minimum and maximum score are 3 and 15 respectively, with higher scores indicating greater sense of belonging.

CONTACTS AND LOCATIONS:
Overall Officials: Devlynne S Ondusko, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared with institutionally IRB approved study team members for data analysis. All other IPD will only be shared in publication in a de-identified, aggregated manner.